CLINICAL TRIAL: NCT06077721
Title: Effect of Milrinone on the Right Ventricular Strain in Cardiac Surgery
Brief Title: Milrinone on Right Ventricular Strain in Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Yop Kim, MD PhD, Professor of Anesthesiology, Konkuk University Medical Center
Other Study IDs: KUH 2023-09-060
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Ischemic Heart Disease; Valvular Heart Disease
Keywords: Milrinone; strain; systolic function
MeSH Terms: conditions — Myocardial Ischemia; Heart Valve Diseases; Sprains and Strains | interventions — Milrinone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Milrinone — giving intravenous milrinone: 50 mcg/kg loading dose by IV push over 10 minutes, then 0.375-0.75 mcg/kg/ min infusion
  Other Names: Milrinone intravenous administration

SUMMARY:
The purpose of this study is to analyze the changes in right ventricular strain before and after milrinone administration in order to find out whether milrinone improves RV systolic performance in patients undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* patient agree and provide written informed consent.
* patient undergoing elective cardiac surgery
* preoperative LV EF>50% (TTE)

Exclusion Criteria:

* preoperative cardiac dysrhythmia
* preoperative IABP
* use of other inotropic agents

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: valvular heart disease, coronary heart disease
Sampling Method: Non-Probability Sample
Enrollment: 41 (Estimated)
Dates: Start 2023-11-03 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
1. Right ventricular strain | 15 min after milrinone administration

SECONDARY OUTCOMES:
Left ventricular strain | 15 min after milrinone administration
Left ventricular ejection fraction | 15 min after milrinone administration

CONTACTS AND LOCATIONS:
Overall Officials: Soi Lee, Study Director — Konkuk University Medical Center
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided